CLINICAL TRIAL: NCT00149565
Title: Hepatocellular Carcinoma Postoperative Adjuvant Therapy Disease Committee of Taiwan Cooperative Oncology Group
Brief Title: Phase Ⅲ Randomized Trial in Postoperative Hepatocellular Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Chang Gung Memorial Hospital (Other); Tri-Service General Hospital (Other); National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); China Medical University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1297
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2004-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

INTERVENTIONS:
Drug: IFN-α2b

SUMMARY:
* OBJECTIVES

1. To investigate whether adjuvant IFN-α therapy can delay or reduce the 2-5 years recurrence rate in curatively resected HCC .
2. To examine whether adjuvant IFN-α therapy can prolong the disease-free survival in curatively resected HCC.
3. To determine the safety and tolerance of adjuvant IFN-α therapy in postoperative HCC with or without cirrhosis.
4. To investigate the change of activity of HBV and HCV in postoperative HCC patients with adjuvant IFN-α therapy.
5. To correlate the changes of viral status with the clinical outcome in post-operative HCC patients with adjuvant IFN-α therapy.

DETAILED DESCRIPTION:
1. TREATMENT PLAN

   1.1 Eligible patients are randomized to receive adjuvant IFN-α for 53 wks or 1.2 Administration of IFN-α 1.21 IFN-α will be started after randomization. 1.22 IFN-α will be administered by subcutaneous injection at the bed time. 1.23 Escalation of IFN-α dosage. 1.231 During the first 2 days, 1 x 106 u/day will be given. 1.232 If tolerable, the dose of IFN-α will be escalated to 3 x 106 u/day in days 3 and 4, and to 5 x 106 u/day at day 5.

   1.24 After dose escalation, IFN-α 5 x 106 u/day will be given in the following ways 1.241 induction therapy: 5 times per week for the first 4 weeks, followed by 1.242 maintenance therapy: 3 times per weeks for additional 48 weeks. 1.25 Modification of IFN-α dosage 1.251 In the presence of any moderate adverse events (as listing in Appendix II) it required a dose reduction to 3 x 106 u/day.

   1.2511 If any moderate adverse events occur at the 3 x 106 u/day level, the patients will be withdraw from the study; 1.252 In the presence of any severe adverse events (as listing in Appendix II), it requires immediate discontinuation of therapy; 1.2521 IFN-α will be discontinued until a return to baseline or moderate toxicity. Then IFN-α will be reinstituted at the dose level of 3 x 106 u/day; 1.2522 If moderate or severe adverse events occur at the 3 x 106 u/day level, the patients will be withdraw from the study.

   1.253 Flare-up of hepatitis activity, as manifested by increment of serum transaminase per se is not an indication for dose modification; 1.254 If symptoms/signs (S/S) of hepatic decompensation occur after the presence of ALT flare-up during IFN-α therapy, the drug will be held.

   1.2541 The presence of two of following five criteria is considered as evidence of hepatic decompensation: 1.25411 Presence of ascites; 1.25412 Presence of hepatic encephalopathy; 1.25413 hypoalbuminemia with serum albumin < 3 g/dl; 1.25414 hyperbilirubinemia with serum bilirubin > 3 mg/dl; 1.25415 Prolongation of prothrombin time with PT > 2 sec above base-line. 1.2542 Serial workup have to be taken to rule out the presence of other predisposing factor (such as spontaneous bacterial peritonitis, constipation, electrolyte imbalance,...ect) to cause the S/S of hepatic decompensation. If any, start specific treatment.

   1.2543 If S/S of hepatic decompensation recovered with a return of serum ALT to ≦1.5 times upper limit of normal range, IFN-α will be restarted at the level of 3 x 106 u/day and escalated to 5 x 106 u/day within 1 week.

   1.2544 If S/S of hepatic decompensation recovered with persistent elevation of serum ALT > 1.5 times upper limit of normal range, IFN-α will be given and maintained at the level 3 x 106 u/day 3 times per week.

   1.2545 After excluding other specific etiologies and S/S of hepatic decompensation persist longer than 4 weeks, patients will be withdrawn from the study.

   1.2546 Recurrent episodes of hepatic decompensation will be considered as severe adverse events and managed as listing in section 5.252.

   1.255 If symptoms/signs (S/S) of hepatic decompensation occur in the absence of ALT flare-up, the patients will be managed as listing in section 5.252.

   1.256 In the presence of severe bacterial infection such as: bacterial peritonitis, bacterial pneumonia, and .. etc., IFN-a will be held until resolution of infection after adequate antibiotics therapy. Then the patients will be managed as listing in section 5.252.

   1.26 Before IFN-α, if necessary patients will be pretreated with acetaminophen 500 - 1,000 mg, q 6 hours for 4 doses, started 12 hours before IFN-α administration to alleviate the associated flu-like symptoms.

   1.3 Adverse Drug Reaction (ADR) Reports 1.31 Any life threatening and/or unexpected and serious (grade 3 or 4) toxicity will be reported within 48 hours to the principal investigator: Li-Tzong Chen M.D. Cancer Clinical Research Center, National Health Research Institutes, A191 Ward Veteran General Hospital Taipei, 201, Shih-Pai Road, Sec 2, Taipei 112, Taiwan Tel:886-2-8712121-2737; Fax: 886-2-8716467; and/or Per-Jei Chen, M.D., Ph.D. Department of Internal Medicine, National Taiwan University Liver Disease Research Center, National Taiwan University Hospital. Tel: 886-2-3970800-7072 Fax: 886-2-3317624. The initial contact should be made by calling the Coordinate Center of TCOG,at 886-2-7852459. A written report will follow within 7 working days.

   1.32 A written report will be submitted within 7 working days describing any life-threatening or lethal (grade 4 or 5) known reactions (except for grade 4 myelosuppression), and any grade 2 or 3 unknown reactions. The address for submitting ADR reports is: Coordinate Center of TCOG, National Health Research Institutes in Biomedical Science, Academia Sinica, Taipei, Taiwan.

   1.33 Above toxicity grading is according to the ECOG toxicity criteria (Appendix III)

   2.0 Evaluation

   The following tests should be performed within 2 weeks before the initiation of therapy ( as the baseline data) and then repeated as request following the initiation of therapy.

   2.1 Physical examination and comprehensive history are recorded bi-weekly during induction period (first month) and monthly during maintenance therapy (for one year). After first year, patients will be followed bi-monthly. After 6 years , patients will be followed 3 monthly.

   2.2 Complete blood count and liver functional tests (bilirubin direct/indirect, AST/ALT and alkaline phosphatase/gGT albumin AC sugar) will be checked bi-weekly during induction period (first month) and monthly during maintenance therapy (for one year). After first year, patients will be followed bi-monthly. After 6 years, patients will be followed 3 monthly..

   2.3 Chest PA every 4 months for one year and then every 6 months. 2.4 ECG for those with history of cardiac disease at time of symptom recurrence.

   2.5 a-fetoprotein will be checked monthly for one year and then bi-monthly. After 6 years, patients will be followed 3 monthly.

   2.6 Abdominal sonography every 2 months. After 6 years, patients will be followed 3 monthly.

   2.7 Abdominal computed tomography performed every 12 months or whenever abdominal sonography shows suspicious recurrent lesions.

   2.8 Any suspicious lesion found on abdominal sonography and/or computed tomography should undergo angiography and sono-guided biopsy for histological examination.

   2.9 UGI endoscopy at the time of UGI bleeding or dyspepsia. [CANCEAL] 2.91 Preoperative endoscopy is acceptable as the base-line data. [CANCEAL] 2.10 Bone scan at the time of symptoms suggest the occurrence of bony metastases.

   2.11 Serum for HBV and HCV status study collected bi-monthly. 2.12 HBeAg and anti-HBe will be checked every 4 months in those with HBeAg(+). After 6 years, patients will be followed 6 monthly.

   2.13 HBsAg will be checked every 6 months in those with HBsAg(+).

   3.0 Off-study Criteria 3.1 Development of a serious medical condition which makes administration of IFN-α life threatening.

   3.11 Patients present with S/S of hepatic decompensation should be managed as list in sections 5.2544 and 5.2545.

   3.12 as those listed in 5.2511 and 5.2522. 3.2 Occurrence of tumor recurrence. 3.3 Non-compliance by a patient with protocol requirement. 3.4 Patient refusal further therapy. 3.5 Patient death. 3.6 Interruption of IFN-α therapy >4 weeks

   4.0 Statistical Consideration 4.1 Sample size Review of literatures showed that the 2-year survival rate of post-operative HCC was 25% to 60% [7-14]. We estimate that adjuvant IFN-α can improve the 2-year survival rate from 50% to 70%. According to the methods of Casagrande et al.[129], to give a 90% power for detecting the increase of 20% for a two-sided statistical significance test, 134 patients for each of the two treatment arms are needed. 4.2 Randomization Patients are stratified into two strata : one with HBsAg(+),another with HBsAg(-) but with anti-HCV(+). Randomization of patients into control or treatment group is taken within each stratum. Balanced block sizes of two strata for randomization are different. 4.3 Analysis 4.31 The primary objectives are as follows: 4.311 To determine if adjuvant IFN-α can reduce or delay the occurrence in curatively resected HCC. 4.312 To determine if adjuvant IFN-α prolong disease-free survival (DFS) and/or overall survival (OS) in curatively resected HCC. 4.313 To determine the safety and tolerance of IFN-αin post-operative H.C.C patients. 4.314 To evaluate the anti-viral activity of IFN-α in post-operative HCC patients. 4.32 DFS and OS are computed from the date of randomization. 4.321 In analysis of DFS, patients died without disease recurrence will be censored for recurrence at the date of death. 4.322 In analysis of OS, an event is defined as death from any cause. 4.323 The survival distributions of DFS and OS will be estimated by the Kaplan and Meier method [130]. 4 4.324 Statistical comparisons of DFS and OS between the two treatment arms will be performed with the log-rank statistic [131]. 4.325 Cox proportional hazards model [132] will be used to assess the importance of potential prognostic factors, as well as to test the significance of treatment when adjusting for factors. 4.33 Tumor size, Liver inflammation, viral status such as HBsAg. anti- HCVand
   * Patient's Specific Factor:

   Performance status Age Sex Family history of HCC and liver diseases. Esophageal varices Prior Hx of esophageal varices bleeding Serum ALT (SGPT) level Serum albumin level Pre-operative serum α-FP level
   * Underlying Liver Disease's Specific Factors:

   HBsAg (by RIA) HBeAg (by RIA) anti-HBc anti-δ antibody anti-HCV antibody Severity of underlying liver disease in nontumor portion Concurrent management of esophageal varices
   * Tumor's Specific Factors:

   Presence of capsule Tumor type Venous invasion Tumor size (the largest in multiple lesions) Histological grading will be treated as potential prognostic factors.

   4.4 Interim Analysis The interim analyses will be conducted according to the alpha spending function approach proposed by DeMets and Lan (1994) which provides flexibility about the time for interim analysis. The a1 spending function, which generates the approximate O'Brien-Fleming boundaries (O'Brien and Fleming, 1979), will be used for a conservation termination at the early stage of the study. In addition, the method of B-value developed by Lan and Wittes (1988), Li (1998) will be used to monitor the data and to compute the conditional probability of detecting either a positive or negative treatment effect at the scheduled end of the study given the present status. The primary efficacy endpoint for the interim analyses is the time to occurrence of second primary tumors. The toxicity will be monitored constantly throughout the study. The conduct of interim analyses and dissemination of the results of the interim analysis will follow the TCOG Data and Safety Monitoring guidelines for confidentiality. The TCOG Data and Safety Monitoring Committee will review the results of interim analyses for a possible early termination of the trial.

ELIGIBILITY:
* Inclusion Criteria:

  1. Histologically proven hepatocellular carcinoma.
  2. HCC underwent curative resection within 6 weeks before registration.
  3. Grossly, the resection margin should be > 1 cm.
  4. Patients must be younger than 70 year-old.
  5. Patients must have a performance status of ECOG score < 2.
  6. Patients must have adequate liver reservation and adequate hemogram.
  7. Pugh-Child's Score < 7.
  8. The serum total bilirubin level are < 2 mg/dl.
  9. The prothrombin times are < 3 sec above normal control.
  10. The platelet are > 10 x 104 / mm3.
  11. The WBC are > 3,000 / mm3.
  12. Patient must have serum creatinine < 1.5 mg/dl
  13. Cardiac function with NYHA classification < Grade II
  14. Known HBV or HCV status.
  15. Signed informed consent.
* Exclusion Criteria:

  1. Patients who have non-curative resection are not eligible.
  2. Resected HCCs with histologically positive margins are not eligible.
  3. HCCs with radiological evidence of portal vein thrombus are not eligible.
  4. Patients with other systemic diseases which required concurrent usage of glucocorticosteroid or immunosuppressant agent(s) are not eligible.
  5. Patients with advanced second primary malignancy are not eligible.
  6. Patients with pregnacy or breast-feeding are not eligible.
  7. Patients with severe cardiopulmonary diseases are not eligible.
  8. Patients with clinically significant psychiatric disorder are not eligible.
  9. Patients who had antineoplastic chemotherapeutic or immuno-therapeutic drugs or corticosteroids within 6 weeks of commencing the protocol are not eligible.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 268
Dates: Start 1997-10; Study Completion 2005-07

PRIMARY OUTCOMES:
134 patients for each of the two treatment arms are needed.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, Ph.D., Study Chair — Hepatocellular Carcinoma Postoperative Adjuvant Therapy Disease Committee of TCOG; Pei-Jer Chen, Ph.D., Study Chair — Hepatocellular Carcinoma Postoperative Adjuvant Therapy Disease Committee of TCOG
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Derived] Chen LT, Chen MF, Li LA, Lee PH, Jeng LB, Lin DY, Wu CC, Mok KT, Chen CL, Lee WC, Chau GY, Chen YS, Lui WY, Hsiao CF, Whang-Peng J, Chen PJ; Disease Committee of Adjuvant Therapy for Postoperative Hepatocellular Carcinoma, Taiwan Cooperative Oncology Group, National Health Research Institutes, Zhunan, Taiwan. Long-term results of a randomized, observation-controlled, phase III trial of adjuvant interferon Alfa-2b in hepatocellular carcinoma after curative resection. Ann Surg. 2012 Jan;255(1):8-17. doi: 10.1097/SLA.0b013e3182363ff9. PMID 22104564